CLINICAL TRIAL: NCT07185581
Title: Evaluation of Small Airway Function During COPD Exacerbation and Recovery Using Impulse Oscillometry (IOS) Device
Brief Title: Impulse Oscillometry in COPD Exacerbation
Status: Completed | Type: Observational
Sponsor: Deniz Bilici (Other)
Responsible Party: Sponsor-Investigator, Deniz Bilici, md, Istanbul Medeniyet University
Organization: Istanbul Medeniyet University (Other)
Other Study IDs: 20.12.2023; 2023/0971
Record Dates: First submitted 2025-09-04; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: COPD Exacerbation; COPD
Keywords: copd; exacerbation; ios; small airway
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- mild exacerbations: Patients were divided into two groups: mild exacerbations (group 1) and moderate and severe exacerbations (group 2) based on ROME criteria.
  Interventions: Diagnostic Test: Impulse Oscillometry
- moderate and severe exacerbations: Patients were divided into two groups: mild exacerbations (group 1) and moderate and severe exacerbations (group 2) based on ROME criteria.
  Interventions: Diagnostic Test: Impulse Oscillometry

INTERVENTIONS:
Diagnostic Test: Impulse Oscillometry — Impulse Oscillometry (IOS) is a simple, non-invasive, effort-independent method that uses sound waves to detect airway changes quickly. It only requires the patient to breathe normally to assess lung function by measuring both resistance and reactance of the airways. 6,7 These features of IOS suggest it may be a useful test for assessing patient respiratory function during exacerbation periods when airway resistance, airflow limitation, and respiratory muscle weakness further impair breathing.
  Other Names: ios

SUMMARY:
This study aimed to evaluate small airway function during ECOPD and recovery periods using IOS. In this prospective single-center study, patients with ECOPD underwent evaluation of their pulmonary functions using IOS and spirometry during exacerbation and recovery (6-12 weeks after exacerbation). The patients were divided into two groups: mild exacerbations and (moderate and severe) exacerbations based on ROME criteria.A total of 41 patients were initially enrolled, with 38 completing the study. This study reveals that IOS can be easily used in ECOPD, and IOS parameters that reflect small airways (R5-R20, AX, and Fres) are correlated with FEV1% and the severity of dyspnea. Additionally, IOS parameters significantly improve during recovery, except for R20. Further research is necessary on its application in the functional assessment of patients with COPD exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* patients who were consecutively admitted to the emergency department or pulmonology outpatient clinic of our hospital with a diagnosis of ECOPD, as defined by the GOLD 2023 Report

Exclusion Criteria:

* Patients diagnosed with pneumonia, pulmonary embolism, heart failure, pleural effusion, or pneumothorax were excluded.
* Patients who were unable to perform spirometry during exacerbation or had a forced expiratory volume in one second (FEV1) to forced vital capacity (FVC) ratio of ≥ 0.70 were also excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 41 patients who were consecutively admitted to the emergency department or pulmonology outpatient clinic of our hospital with a diagnosis of ECOPD, as defined by the GOLD 2023 Report 1 , were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Physiological parameter of IOS in COPD exacerbation period | from baseline
  We investigated descriptive parameters of impulse oscillometry during copd exacerbation period to use in clinical setting in the future.
  The parameters for assessing airway resistance, including resistance at 5 Hz (R5), which indicates total airway resistance; resistance at 20 Hz (R20), representing the resistance of large airways; and the difference between resistance at 5 Hz and 20 Hz ( R5-R20 ). The parameters that assess reactance are X5, which measures peripheral elastic resistance at 5 Hz; AX, the area under the reactance curve between 5 Hz and the resonant frequency, reflecting the elastic properties of the lung; and Fres, the oscillation frequency at which reactance is zero.
  In the exacerbation of copd period FEV1% was correlated with all IOS parameters except R20, and BORG was correlated with IOS parameters except R20 and X5. Furthermore, IOS parameters reflecting the small airways (R5-R20, X5, AX, Fres) also showed strong intercorrelations.

SECONDARY OUTCOMES:
Comparison of parameter of IOS in COPD exacerbation period to stable period (approximately 6 weeks later) | 6 weeks later from the baseline
  Thirty-eight patients were re-evaluated during the recovery period. Significant improvements were observed in R5, R5-R20, AX, and Fres during recovery. No differences were observed in IOS parameters based on the severity of exacerbation.
Comparison and correlations of IOS and pulmonary function test parameters in recovery period of COPD patient | 6 weeks later from the baseline
  We investigated correlation of IOS parameters such as R5, R5-R20, X5, AX, and Fres with pulmonary function test paramteres such as FEV1%, FVC%, FEV1/FVC We measured these parameters both in exacerbation and recovery periods of same patients and compared the results of two tests measurements

CONTACTS AND LOCATIONS:
Overall Officials: Esma Seda Akalın, MD, Principal Investigator — Istanbul Medeniyet University; Deniz Koçak, Research Assistant, Principal Investigator — Istanbul Medeniyet University; Elif Hazal Karadağ, Research Assistant, Principal Investigator — Istanbul Medeniyet University; Burcu Arpınar Yiğitbaş, Associate professor:, Principal Investigator — Istanbul Medeniyet University; Deniz Bilici, MD, Principal Investigator — Istanbul Medeniyet University; Handan Ankaralı, Professor, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
All IPD used in the results publication

REFERENCES:
- [Result] Anderson WJ, Lipworth BJ. Relationships between impulse oscillometry, spirometry and dyspnoea in COPD. J R Coll Physicians Edinb. 2012 Jun;42(2):111-5. doi: 10.4997/JRCPE.2012.204. PMID 22693693
- [Result] Haruna A, Oga T, Muro S, Ohara T, Sato S, Marumo S, Kinose D, Terada K, Nishioka M, Ogawa E, Hoshino Y, Hirai T, Chin K, Mishima M. Relationship between peripheral airway function and patient-reported outcomes in COPD: a cross-sectional study. BMC Pulm Med. 2010 Mar 7;10:10. doi: 10.1186/1471-2466-10-10. PMID 20205936
- [Result] Huang Y, Zhang X, Wang J, Bao W, Lv C, Zhang Y, Tian X, Zhou Y, Zhang M. Role of impulse oscillometry in chronic obstructive pulmonary disease and asthma-chronic obstructive pulmonary disease overlap. Clin Transl Allergy. 2025 Apr;15(4):e70057. doi: 10.1002/clt2.70057. PMID 40261129
- [Result] Gao L, Wang H, Wu Y, Wang T, Xiong S, Qiu R, Zhou H, Liu L, Jia H, Qin J, Xu D, Shen Y, Chen L, Wen FQ. Diagnostic value of impulse oscillometry in chronic obstructive pulmonary disease: a multicentre, retrospective, observational study. BMJ Open. 2024 Oct 8;14(10):e087687. doi: 10.1136/bmjopen-2024-087687. PMID 39384230
- [Result] Wei X, Shi Z, Cui Y, Mi J, Ma Z, Ren J, Li J, Xu S, Guo Y. Impulse oscillometry system as an alternative diagnostic method for chronic obstructive pulmonary disease. Medicine (Baltimore). 2017 Nov;96(46):e8543. doi: 10.1097/MD.0000000000008543. PMID 29145259
- [Result] Lu L, Peng J, Wu F, Yang H, Zheng Y, Deng Z, Zhao N, Dai C, Xiao S, Wen X, Xu J, Wu X, Zhou K, Ran P, Zhou Y. Clinical characteristics of airway impairment assessed by impulse oscillometry in patients with chronic obstructive pulmonary disease: findings from the ECOPD study in China. BMC Pulm Med. 2023 Feb 3;23(1):52. doi: 10.1186/s12890-023-02311-z. PMID 36737731
- [Result] Zheng S, Hu Y, Chen Z, Wang M, Liao W. Predicting asthma exacerbation by impulse oscillometry evaluation of small airway function and fractional exhaled nitric oxide in preschool children. Pediatr Pulmonol. 2020 Jul;55(7):1601-1607. doi: 10.1002/ppul.24790. Epub 2020 Apr 30. PMID 32353216
- [Result] Schulze J, Biedebach S, Christmann M, Herrmann E, Voss S, Zielen S. Impulse Oscillometry as a Predictor of Asthma Exacerbations in Young Children. Respiration. 2016;91(2):107-14. doi: 10.1159/000442448. Epub 2016 Jan 13. PMID 26756585
- [Result] Ling Y, Si M, Niu Y, Han Y, Xu Y. The predictive value of impulse oscillometry for asthma exacerbations in childhood: A systematic review and meta-analyses. Pediatr Pulmonol. 2021 Jul;56(7):1850-1856. doi: 10.1002/ppul.25374. Epub 2021 Mar 23. PMID 33756052
- [Result] Park H, Lee HJ, Lee HW, Park TY, Heo EY, Kim DK, Lee JK. Diagnosis and evaluation of small airway disease and COPD using impulse oscillometry. Sci Rep. 2024 Nov 14;14(1):28030. doi: 10.1038/s41598-024-79818-w. PMID 39543228
- [Result] Su ZQ, Guan WJ, Li SY, Ding M, Chen Y, Jiang M, Chen XB, Zhong CH, Tang CL, Zhong NS. Significances of spirometry and impulse oscillometry for detecting small airway disorders assessed with endobronchial optical coherence tomography in COPD. Int J Chron Obstruct Pulmon Dis. 2018 Oct 1;13:3031-3044. doi: 10.2147/COPD.S172639. eCollection 2018. PMID 30319251
- [Result] Duman D, Tasti OF, Merve Tepetam F. Assessment of small airway dysfunction by impulse oscillometry (IOS) in COPD and IPF patients. Eur Rev Med Pharmacol Sci. 2023 Apr;27(7):3033-3044. doi: 10.26355/eurrev_202304_31937. PMID 37070906
- [Result] Williamson PA, Clearie K, Menzies D, Vaidyanathan S, Lipworth BJ. Assessment of small-airways disease using alveolar nitric oxide and impulse oscillometry in asthma and COPD. Lung. 2011 Apr;189(2):121-9. doi: 10.1007/s00408-010-9275-y. Epub 2010 Dec 22. PMID 21174112
- [Result] Yanai M, Sekizawa K, Ohrui T, Sasaki H, Takishima T. Site of airway obstruction in pulmonary disease: direct measurement of intrabronchial pressure. J Appl Physiol (1985). 1992 Mar;72(3):1016-23. doi: 10.1152/jappl.1992.72.3.1016. PMID 1568955
- [Result] Hogg JC, Macklem PT, Thurlbeck WM. Site and nature of airway obstruction in chronic obstructive lung disease. N Engl J Med. 1968 Jun 20;278(25):1355-60. doi: 10.1056/NEJM196806202782501. No abstract available. PMID 5650164
- [Result] Lipworth BJ, Jabbal S. What can we learn about COPD from impulse oscillometry? Respir Med. 2018 Jun;139:106-109. doi: 10.1016/j.rmed.2018.05.004. Epub 2018 May 16. PMID 29857993
- [Result] Xu J, Sun X, Zhu H, Cao Y, Pudasaini B, Yang W, Liu J, Guo J. Long-term variability of impulse oscillometry and spirometry in stable COPD and asthma. Respir Res. 2022 Sep 21;23(1):262. doi: 10.1186/s12931-022-02185-5. PMID 36131305
- [Result] Kolsum U, Borrill Z, Roy K, Starkey C, Vestbo J, Houghton C, Singh D. Impulse oscillometry in COPD: identification of measurements related to airway obstruction, airway conductance and lung volumes. Respir Med. 2009 Jan;103(1):136-43. doi: 10.1016/j.rmed.2008.07.014. Epub 2008 Aug 28. PMID 18760576
- [Result] Crim C, Celli B, Edwards LD, Wouters E, Coxson HO, Tal-Singer R, Calverley PM; ECLIPSE investigators. Respiratory system impedance with impulse oscillometry in healthy and COPD subjects: ECLIPSE baseline results. Respir Med. 2011 Jul;105(7):1069-78. doi: 10.1016/j.rmed.2011.01.010. Epub 2011 Apr 11. PMID 21481577
- [Result] Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. General considerations for lung function testing. Eur Respir J. 2005 Jul;26(1):153-61. doi: 10.1183/09031936.05.00034505. No abstract available. PMID 15994402
- [Result] Oostveen E, MacLeod D, Lorino H, Farre R, Hantos Z, Desager K, Marchal F; ERS Task Force on Respiratory Impedance Measurements. The forced oscillation technique in clinical practice: methodology, recommendations and future developments. Eur Respir J. 2003 Dec;22(6):1026-41. doi: 10.1183/09031936.03.00089403. PMID 14680096
- [Result] Chen Y, Pei Y, Mo W, Wang H. The Relationship Between Serum Inflammatory Markers and Chronic Obstructive Pulmonary Disease in Middle-Aged and Older Adults in the United States: A Cross-Sectional Study Based on NHANES 2013-2018. Int J Chron Obstruct Pulmon Dis. 2025 Aug 13;20:2837-2846. doi: 10.2147/COPD.S534504. eCollection 2025. PMID 40827237
- [Result] Xu Y, Yan Z, Li K, Liu L. The association between systemic immune-inflammation index and chronic obstructive pulmonary disease in adults aged 40 years and above in the United States: a cross-sectional study based on the NHANES 2013-2020. Front Med (Lausanne). 2023 Nov 24;10:1270368. doi: 10.3389/fmed.2023.1270368. eCollection 2023. PMID 38076255
- [Result] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Result] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Result] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201
- [Result] Komarow HD, Myles IA, Uzzaman A, Metcalfe DD. Impulse oscillometry in the evaluation of diseases of the airways in children. Ann Allergy Asthma Immunol. 2011 Mar;106(3):191-9. doi: 10.1016/j.anai.2010.11.011. Epub 2011 Jan 6. PMID 21354020
- [Result] DUBOIS AB, BRODY AW, LEWIS DH, BURGESS BF Jr. Oscillation mechanics of lungs and chest in man. J Appl Physiol. 1956 May;8(6):587-94. doi: 10.1152/jappl.1956.8.6.587. No abstract available. PMID 13331841
- [Result] Global Initiative for Asthma (GINA). Global strategy for asthma management and prevention. http://www.ginasthma.org. Date last updated: August 26 2025. Date last accessed: August 26 2025.
- [Result] Celli BR, Fabbri LM, Aaron SD, Agusti A, Brook R, Criner GJ, Franssen FME, Humbert M, Hurst JR, O'Donnell D, Pantoni L, Papi A, Rodriguez-Roisin R, Sethi S, Torres A, Vogelmeier CF, Wedzicha JA. An Updated Definition and Severity Classification of Chronic Obstructive Pulmonary Disease Exacerbations: The Rome Proposal. Am J Respir Crit Care Med. 2021 Dec 1;204(11):1251-1258. doi: 10.1164/rccm.202108-1819PP. No abstract available. PMID 34570991
- [Result] Vogelmeier CF, Criner GJ, Martinez FJ, Anzueto A, Barnes PJ, Bourbeau J, Celli BR, Chen R, Decramer M, Fabbri LM, Frith P, Halpin DM, Lopez Varela MV, Nishimura M, Roche N, Rodriguez-Roisin R, Sin DD, Singh D, Stockley R, Vestbo J, Wedzicha JA, Agusti A. Global Strategy for the Diagnosis, Management, and Prevention of Chronic Obstructive Lung Disease 2017 Report. GOLD Executive Summary. Am J Respir Crit Care Med. 2017 Mar 1;195(5):557-582. doi: 10.1164/rccm.201701-0218PP. PMID 28128970
- [Result] 1.Agustí A, Celli BR, Criner GJ et al. Global Initiative for Chronic Obstructive Lung Disease 2023 Report: GOLD Executive Summary. Eur Respir J 2023; 61(4):2300239. 2.Wedzicha JA, Seemungal TA. COPD exacerbations: defining their cause and prevention. Lancet 2007; 370(9589): 786-796.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/81/NCT07185581/Prot_SAP_000.pdf